CLINICAL TRIAL: NCT05752786
Title: Evaluation of the Effect of the "Eat Less Meat" One-month Challenge on Meat Consumption Among French University Students
Brief Title: Evaluation of the "Eat Less Meat" One-month Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EIPH0154
Record Dates: First submitted 2023-02-01; First posted 2023-03-03 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Diet, Healthy; Food Habits
Keywords: meat reduction; environmental impact; nutritional quality; diet
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Eat Less Meat" challenge (Experimental): Participants take part in the "Eat Less Meat" challenge
  Interventions: Behavioral: "Eat Less Meat" Challenge
- "Eat Less Meat" challenge later (Other): Participants take part in the "Eat Less Meat" challenge 4 months after the participants in the experimental arm, i.e., after all measures completion
  Interventions: Behavioral: "Eat Less Meat" Challenge

INTERVENTIONS:
Behavioral: "Eat Less Meat" Challenge — Participants will be able to choose their goal for the challenge for one month: (i) no meat, (ii) meat 3 times a week, (iii) meat 6 times a week (which will need to be lower than current consumption). The first day of the challenge, the participants will receive by email a cookbook and a starter kit with advices and motivational tips, then they will receive an email each week with more advices and motivational tips. Participants will be also asked to follow the Instagram account of the challenge during one month where (i) one post will be posted each day, (ii) engaging stories requiring interactions will be posted regularly, (iii) participants can ask their questions to the research team, (iv) participants can interact with each other's. The Instagram posts will cover three main topics: (i) knowledge about meat and its impact on health and environment, (ii) tips for meat-free cooking, (iii) social/contextual pressure to eat meat and how to avoid it.

SUMMARY:
In a context where meat consumption should be dramatically reduced in western countries to improve both population and planet health, the "Eat Less Meat" one-month challenge is a new behavioural intervention that aims (i) to weaken meat consumption habit and (ii) to enhance intrinsic motivation to eat less meat to trigger long-term reduction in meat consumption. The present study focusses on the quantitative evaluation of the effect of this challenge on French university student's meat consumption.

Parallel two-arm randomized controlled trial with repeated measures (online questionnaires) pre-, during- and post-intervention. All the participants will be recruited to take part in the "Eat Less Meat" challenge for one month. Participants in the control group will take part in the challenge 4 months after the participants in the intervention group. Participants in both groups will complete the online questionnaires at the exact same time, i.e., pre-, during- and post-intervention measures will take place before the control group starts the challenge.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 18.5
* University student in 'Bourgogne Franche-Comté'
* Fluent in French
* Available email address
* Available Instagram profile

Exclusion Criteria:

* Vegetarian or vegan or pescetarian
* Pregnant/breastfeeding
* Iron deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Meat consumption at 1 month (during intervention) | 20 minutes, repeated measures (online food frequency questionnaire): baseline and month 1
  Meat daily intake (in grams) will be calculated by summing daily intake for all the items of the food frequency questionnaire that fall into the meat category.
Change from Baseline Meat consumption at 4 months (3 months after intervention) | 20 minutes, repeated measures (online food frequency questionnaire): baseline and month 4
  Meat daily intake (in grams) will be calculated by summing daily intake for all the items of the food frequency questionnaire that fall into the meat category.

SECONDARY OUTCOMES:
Change from Baseline Adherence to the French dietary guidelines at 1 month (during intervention) | 20 minutes, repeated measures (online food frequency questionnaire): baseline and month 1
  Adherence to the French dietary guidelines will be evaluated using the simplified PNNS-GS2. The sPNNS-GS2 builds on the distinction between malus components (less healthy food groups which consumption should be limited, carrying a negative score, i.e., red meat, processed meat, sugary foods, sweet-tasting beverages, alcoholic beverages, salt) and bonus components (healthier food groups carrying a positive score, i.e., fruits and vegetables, nuts, legumes, whole-grain food, milk and dairy products, fish and seafood) reflecting established knowledge on the relationship between food groups consumption and non-communicable disease risk factors. sPNNS-GS2 will computed for each participant (range: -17 to 11.5, with higher scores indicating better adherence to the French dietary guidelines).
Change from Baseline Adherence to the French dietary guidelines at 4 months (3 months after intervention) | 20 minutes, repeated measures (online food frequency questionnaire): baseline and month 4
  Adherence to the French dietary guidelines will be evaluated using the simplified PNNS-GS2. The sPNNS-GS2 builds on the distinction between malus components (less healthy food groups which consumption should be limited, carrying a negative score, i.e., red meat, processed meat, sugary foods, sweet-tasting beverages, alcoholic beverages, salt) and bonus components (healthier food groups carrying a positive score, i.e., fruits and vegetables, nuts, legumes, whole-grain food, milk and dairy products, fish and seafood) reflecting established knowledge on the relationship between food groups consumption and non-communicable disease risk factors. sPNNS-GS2 will computed for each participant (range: -17 to 11.5, with higher scores indicating better adherence to the French dietary guidelines).
Change from Baseline Greenhouse gas emissions at 1 month (during intervention) | 20 minutes, repeated measures (online food frequency questionnaire): baseline and month 1
  Greenhouse gas emissions (GHGEs) will be calculated by multiplying the daily intake of each food item by its associated GHGEs per kg
Change from Baseline Greenhouse gas emissions at 4 months (3 months after intervention) | 20 minutes, repeated measures (online food frequency questionnaire): baseline and month 4
  Greenhouse gas emissions (GHGEs) will be calculated by multiplying the daily intake of each food item by its associated GHGEs per kg
Change from Baseline Meat consumption habit at 1 month (during intervention) | 3 minutes, repeated measures (online Self-Report Habit questionnaire): baseline and month 1
  The Self-Report Habit Index will be computed by averaging ratings for all the 12 individual items from the Self-Report Habit questionnaire. Responses will be reported on a 6-point scale anchored by 'strongly disagree' and 'strongly agree' from 1 to 6. The scores will be coded such that high values indicated strong habits.
Change from Baseline Meat consumption habit at 4 months (3 months after intervention) | 3 minutes, repeated measures (online Self-Report Habit questionnaire): baseline and month 4
  The Self-Report Habit Index will be computed by averaging ratings for all the 12 individual items from the Self-Report Habit questionnaire. Responses will be reported on a 6-point scale anchored by 'strongly disagree' and 'strongly agree' from 1 to 6. The scores will be coded such that high values indicated strong habits.
Change from Baseline Food choice motives at 1 month (during intervention) | 5 minutes, repeated measures (online food choice motives questionnaire): baseline and month 1
  The food choice questionnaire (FCQ) includes 30 items and 10 subscales: health, mood, convenience, sensory appeal, natural content, price, weight control, familiarity, ethical concern and animal welfare. Answers to each item will range from 1 to 4: 1 = Not at all important; 2 = A little important; 3 = Moderately important; 4 = Very important. A score for each motive will be computed by averaging ratings for the three individual items in each of the ten subscales, higher scores indicating higher importance.
Change from Baseline Food choice motives at 4 months (3 months after intervention) | 5 minutes, repeated measures (online food choice motives questionnaire): baseline and month 4
  The food choice questionnaire (FCQ) includes 30 items and 10 subscales: health, mood, convenience, sensory appeal, natural content, price, weight control, familiarity, ethical concern and animal welfare. Answers to each item will range from 1 to 4: 1 = Not at all important; 2 = A little important; 3 = Moderately important; 4 = Very important. A score for each motive will be computed by averaging ratings for the three individual items in each of the ten subscales, higher scores indicating higher importance.

CONTACTS AND LOCATIONS:
Overall Officials: Lucile Marty, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
Share on Open Science Framework
Supporting Information: Study Protocol, SAP
Time Frame: Before data collection, indefinitely
Access Criteria: Open website
URL: https://osf.io/3gts8/

REFERENCES:
- [Derived] Marty L, Biehlmann M, Louveau A, Poquet D, Robinson E. The "Eat Less Meat" one-month challenge: a randomized controlled trial of a meat reduction pledge intervention among French university students. Int J Behav Nutr Phys Act. 2025 Oct 27;22(1):131. doi: 10.1186/s12966-025-01831-7. PMID 41146183
- Available data/document: Study Protocol — https://osf.io/3gts8/
- Available data/document: Statistical Analysis Plan — https://osf.io/3gts8/
- Available data/document: Individual Participant Data Set — https://osf.io/3gts8/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05752786/Prot_SAP_000.pdf